CLINICAL TRIAL: NCT00931944
Title: An Open-Label, Safety and Tolerability, Study Evaluating KNS-760704 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Open-Label, Safety and Tolerability Extension Study of KNS-760704 in Amyotrophic Lateral Sclerosis (ALS) (CL211)
Acronym: CL211
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNS-760704-CL211
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig; Lou Gehrig's; Lou Gehrig's disease; Motor Neuron Disease; Nervous System Diseases; KNS-760704; RTPB
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Nervous System Diseases | interventions — Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KNS-760704 300 mg/day (Experimental): Open-label KNS-760704 (150 mg Q12H)
  Interventions: Drug: KNS-760704

INTERVENTIONS:
Drug: KNS-760704 — 150 mg Q12H KNS-760704 given orally (300 mg total daily dose)
  Other Names: dexpramipexole

SUMMARY:
This is an open-label, multi-center study designed to extend the evaluation of the safety, tolerability, and clinical effects of oral administration of KNS-760704 in patients with ALS.

DETAILED DESCRIPTION:
Patients who complete the Part 2 Week 28 visit in study KNS-760704-CL201 and patients with ALS who were actively receiving RTPB [(6R)-4,5,6,7-tetrahydro-N6-propyl-2,6-benzothiazolediamine dihydro-chloride monohydrate] under Research IND #60,948 were eligible to participate in this study.

Eligible patients received 1 tablet of KNS-760704 (150 mg) every 12 hours (Q12H) (300 mg total daily dose) for up to 180 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided signed informed consent for this trial before the commencement of any study-related procedure
2. Patient is actively participating in Knopp Protocol KNS-760704-CL201 and has completed the Part 2 Week 28 visit in that study or patient is actively receiving RTPB under Research IND #60,948

Exclusion Criteria:

1. Patient did not participate in Knopp Protocol KNS-760704-CL201 or patient did not receive RTPB under Research IND #60,948.
2. Patient discontinued from KNS-760704-CL201 for any reason other than enrollment into this study (applies to patients enrolled in KNS-760704-CL201 only)
3. Patient was not taking RTPB under Research IND #60,948 prior to April 30, 2009 (applies to patients enrolled under Research IND #60,948 only)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, M.D., MSc, Principal Investigator — NeuroClinical Trials Unit (Massachusetts General Hospital)
Locations (19):
- United States (19):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA, Dept. of Neurology - Neuromuscular/ALS Research Center, Los Angeles, California
  - The Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusettes General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Columbia University, Lou Gehrig MDA/ALS Research Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College Of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Sciences Center of San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 300 mg Per Day: KNS-760704 (dexpramipexole) - 150 mg BID
Period: Overall Study
Arm/Group | 300 mg Per Day
Started | 74
Completed | 19
Not Completed | 55
Not completed — Adverse Event | 4
Not completed — W/D Consent (due to ALS progression)) | 19
Not completed — Withdrawal Consent (due to other) | 2
Not completed — Death | 28
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Safety Population was defined as all subjects who received at least 1 dose of study treatment during the study.
Arm/Group | 300 mg Per Day
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.14)
Age, Customized [Count of Participants; unit: Participants]
  <=50 | 24
  51-65 | 30
  >65 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 72
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Potentially Clinically Significant Hematology Results
Description: Number of Participants with Potentially Clinically Significant Hematology Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: 180 weeks
Population: Number of subjects evaluated is the number of subjects who had a baseline assessment and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 74
Participants
  WBC (<3.0 x 10^9/L): number analyzed (Participants) | 72
  WBC (<3.0 x 10^9/L) | 5
  WBC (>=16.0 x 10^9/L): number analyzed (Participants) | 72
  WBC (>=16.0 x 10^9/L) | 2
  Neutrophils (<1.5 x 10^9/L): number analyzed (Participants) | 71
  Neutrophils (<1.5 x 10^9/L) | 3
  Neutrophils (>13.5 x 10^9/L): number analyzed (Participants) | 71
  Neutrophils (>13.5 x 10^9/L) | 4

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Liver Enzyme Abnormalities
Description: Number of participants with potentially clinically significant liver enzyme abnormalities for the safety population are presented. Percentages are based on the number of patients with at least one non-missing, post-baseline value for each parameter.
Time Frame: 180 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 74
Participants
  Alkaline phosphatase >2.5 times ULN (upper limit of the 'normal' reference range): number analyzed (Participants) | 72
  Alkaline phosphatase >2.5 times ULN (upper limit of the 'normal' reference range) | 1
  ALT >3 times ULN: number analyzed (Participants) | 72
  ALT >3 times ULN | 5
  AST >3 times ULN: number analyzed (Participants) | 72
  AST >3 times ULN | 2
  Total Bilirubin >1.5 times ULN: number analyzed (Participants) | 72
  Total Bilirubin >1.5 times ULN | 3
  Creatinine >1.5 times ULN: number analyzed (Participants) | 64
  Creatinine >1.5 times ULN | 0
  ALT or AST >3 times ULN and total bilirubin >2 times ULN (Hy's Law): number analyzed (Participants) | 72
  ALT or AST >3 times ULN and total bilirubin >2 times ULN (Hy's Law) | 0

3. Primary Outcome: Number of Participants With Potentially Clinically ECG Abnormalities
Description: Number of participants with potentially clinically significant ECG abnormalities for the safety population are presented. Percentages are based on the number of patients in the safety population who had at least one non-missing, post-baseline value.
Time Frame: 180 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 74
Participants
  Axis - LEFT AXIS DEVIATION: number analyzed (Participants) | 68
  Axis - LEFT AXIS DEVIATION | 5
  Axis - RIGHT AXIS DEVIATION: number analyzed (Participants) | 68
  Axis - RIGHT AXIS DEVIATION | 1
  Conduction - LEFT ANTERIOR HEMIBLOCK: number analyzed (Participants) | 56
  Conduction - LEFT ANTERIOR HEMIBLOCK | 2
  Conduction - RSR' SUGGESTS RIGHT VENTRICULAR CONDUCTION DELAY: number analyzed (Participants) | 56
  Conduction - RSR' SUGGESTS RIGHT VENTRICULAR CONDUCTION DELAY | 3
  Conduction - SHORT P-R INTERVAL: number analyzed (Participants) | 56
  Conduction - SHORT P-R INTERVAL | 3
  Morphology - LEFT ATRIAL ENLARGEMENT: number analyzed (Participants) | 64
  Morphology - LEFT ATRIAL ENLARGEMENT | 2
  Morphology - LEFT VENTRICULAR HYPERTROPHY BY VOLTAGE CRITERIA ONLY: number analyzed (Participants) | 64
  Morphology - LEFT VENTRICULAR HYPERTROPHY BY VOLTAGE CRITERIA ONLY | 2
  Morphology - LEFT VENTRICULAR HYPERTROPHY WITH REPOLARIZATION ABNORMALITIES: number analyzed (Participants) | 64
  Morphology - LEFT VENTRICULAR HYPERTROPHY WITH REPOLARIZATION ABNORMALITIES | 1
  Morphology - POSSIBLE RIGHT VENTRICULAR HYPERTROPHY: number analyzed (Participants) | 64
  Morphology - POSSIBLE RIGHT VENTRICULAR HYPERTROPHY | 1
  Morphology - RIGHT VENTRICULAR HYPERTROPHY: number analyzed (Participants) | 64
  Morphology - RIGHT VENTRICULAR HYPERTROPHY | 1
  Myocardial Ischemia/Infarction - ANTEROSEPTAL MYOCARDIAL INFARCTION - AGE UNDETERMINED: number analyzed (Participants) | 66
  Myocardial Ischemia/Infarction - ANTEROSEPTAL MYOCARDIAL INFARCTION - AGE UNDETERMINED | 1
  Myocardial Ischemia/Infarction - CANNOT RULE OUT POSSIBLE MYOCARDIAL INFARCTION (INFERIOR): number analyzed (Participants) | 66
  Myocardial Ischemia/Infarction - CANNOT RULE OUT POSSIBLE MYOCARDIAL INFARCTION (INFERIOR) | 1
  Myocardial Isch/Infar. CANNOT RULE OUT POSSIBLE MYOCARDIAL INFARCTION MAY BE IMPROPER LEAD POSITIONS: number analyzed (Participants) | 66
  Myocardial Isch/Infar. CANNOT RULE OUT POSSIBLE MYOCARDIAL INFARCTION MAY BE IMPROPER LEAD POSITIONS | 1
  Myocardial Ischemia/Infarction - INFERIOR MYOCARDIAL INFARCTION - AGE UNDETERMINED: number analyzed (Participants) | 66
  Myocardial Ischemia/Infarction - INFERIOR MYOCARDIAL INFARCTION - AGE UNDETERMINED | 1
  Myocardial Ischemia/Infarction - OLD INFERIOR MYOCARDIAL INFARCTION: number analyzed (Participants) | 66
  Myocardial Ischemia/Infarction - OLD INFERIOR MYOCARDIAL INFARCTION | 1
  Other - POOR PRECORDIAL R WAVE PROGRESSION. POSSIBLE IMPROPER PLACEMENT OF V LEADS.: number analyzed (Participants) | 72
  Other - POOR PRECORDIAL R WAVE PROGRESSION. POSSIBLE IMPROPER PLACEMENT OF V LEADS. | 1
  Other - POOR R WAVE PROGRESSION, PRECORDIAL LEADS: number analyzed (Participants) | 72
  Other - POOR R WAVE PROGRESSION, PRECORDIAL LEADS | 3
  QT Interval - QTCB BORDERLINE PROLONGED: number analyzed (Participants) | 70
  QT Interval - QTCB BORDERLINE PROLONGED | 9
  Rhythm - ATRIAL FLUTTER WITH 3:1 VENTRICULAR RESPONSE: number analyzed (Participants) | 57
  Rhythm - ATRIAL FLUTTER WITH 3:1 VENTRICULAR RESPONSE | 1
  Rhythm - FREQUENT VENTRICULAR PREMATURE BEATS: number analyzed (Participants) | 57
  Rhythm - FREQUENT VENTRICULAR PREMATURE BEATS | 1
  Rhythm - RARE VENTRICULAR PREMATURE BEATS: number analyzed (Participants) | 57
  Rhythm - RARE VENTRICULAR PREMATURE BEATS | 1
  Rhythm - SINUS BRADYCARDIA: number analyzed (Participants) | 57
  Rhythm - SINUS BRADYCARDIA | 2
  Rhythm - SINUS TACHYCARDIA: number analyzed (Participants) | 57
  Rhythm - SINUS TACHYCARDIA | 25
  Rhythm - UNUSUAL P AXIS, POSSIBLE ECTOPIC ATRIAL RHYTHM: number analyzed (Participants) | 57
  Rhythm - UNUSUAL P AXIS, POSSIBLE ECTOPIC ATRIAL RHYTHM | 1
  Rhythm - VENTRICULAR PREMATURE BEATS: number analyzed (Participants) | 57
  Rhythm - VENTRICULAR PREMATURE BEATS | 1
  ST-T Wave - COUNTERCLOCKWISE ROTATION: number analyzed (Participants) | 61
  ST-T Wave - COUNTERCLOCKWISE ROTATION | 1
  ST-T Wave - EARLY REPOLARIZATION: number analyzed (Participants) | 61
  ST-T Wave - EARLY REPOLARIZATION | 1
  ST-T Wave - NON-SPECIFIC ST ABNORMALITY: number analyzed (Participants) | 61
  ST-T Wave - NON-SPECIFIC ST ABNORMALITY | 2
  ST-T Wave - NON-SPECIFIC ST AND T WAVE ABNORMALITY: number analyzed (Participants) | 61
  ST-T Wave - NON-SPECIFIC ST AND T WAVE ABNORMALITY | 1
  ST-T Wave - NON-SPECIFIC T WAVE ABNORMALITY: number analyzed (Participants) | 61
  ST-T Wave - NON-SPECIFIC T WAVE ABNORMALITY | 14

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Abnormalities
Description: Number of participants with potentially clinically significant vital sign abnormalities for the safety population are presented. Percentages are based on the number of patients with at least one non-missing, post-baseline value for each parameter.
Time Frame: 180 weeks
Population: Number of subjects evaluated is the number of subjects in the Safety Population who had a baseline assessment and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 74
Participants
  Temperature - >38 degree C. post-baseline and an increase from baseline of at least 1 degree Celsius: number analyzed (Participants) | 72
  Temperature - >38 degree C. post-baseline and an increase from baseline of at least 1 degree Celsius | 4
  Pulse Rate - >120 bpm post-baseline or an increase from baseline of >20 bpm: number analyzed (Participants) | 72
  Pulse Rate - >120 bpm post-baseline or an increase from baseline of >20 bpm | 26
  Pulse Rate - >120 bpm post-baseline and an increase from baseline of >20 bpm: number analyzed (Participants) | 72
  Pulse Rate - >120 bpm post-baseline and an increase from baseline of >20 bpm | 1
  Pulse Rate - <50 bpm post-baseline or a decrease from baseline of >20 bpm: number analyzed (Participants) | 72
  Pulse Rate - <50 bpm post-baseline or a decrease from baseline of >20 bpm | 9
  Pulse Rate - <50 bpm post-baseline and a decrease from baseline of >20 bpm: number analyzed (Participants) | 72
  Pulse Rate - <50 bpm post-baseline and a decrease from baseline of >20 bpm | 0
  Systolic Blood Pressure - >180 mmHg post-baseline or an increase from baseline of >40 mmHg: number analyzed (Participants) | 72
  Systolic Blood Pressure - >180 mmHg post-baseline or an increase from baseline of >40 mmHg | 3
  Systolic Blood Pressure - >180 mmHg post-baseline and an increase from baseline of >40 mmHg: number analyzed (Participants) | 72
  Systolic Blood Pressure - >180 mmHg post-baseline and an increase from baseline of >40 mmHg | 1
  Systolic Blood Pressure - <90 mmHg post-baseline or a decrease from baseline of >30 mmHg: number analyzed (Participants) | 72
  Systolic Blood Pressure - <90 mmHg post-baseline or a decrease from baseline of >30 mmHg | 11
  Systolic Blood Pressure - <90 mmHg post-baseline and a decrease from baseline of >30 mmHg: number analyzed (Participants) | 72
  Systolic Blood Pressure - <90 mmHg post-baseline and a decrease from baseline of >30 mmHg | 1
  Diastolic Blood Pressure - >105 mmHg post-baseline or an increase from baseline of >30 mmHg: number analyzed (Participants) | 72
  Diastolic Blood Pressure - >105 mmHg post-baseline or an increase from baseline of >30 mmHg | 4
  Diastolic Blood Pressure - >105 mmHg post-baseline and an increase from baseline of >30 mmHg: number analyzed (Participants) | 72
  Diastolic Blood Pressure - >105 mmHg post-baseline and an increase from baseline of >30 mmHg | 0
  Diastolic Blood Pressure - <50 mmHg post-baseline or a decrease from baseline of >20 mmHg: number analyzed (Participants) | 72
  Diastolic Blood Pressure - <50 mmHg post-baseline or a decrease from baseline of >20 mmHg | 13
  Diastolic Blood Pressure - <50 mmHg post-baseline and a decrease from baseline of >20 mmHg: number analyzed (Participants) | 72
  Diastolic Blood Pressure - <50 mmHg post-baseline and a decrease from baseline of >20 mmHg | 0
  Weight - Increase from baseline of >7%: number analyzed (Participants) | 72
  Weight - Increase from baseline of >7% | 4
  Weight - Decrease from baseline of >7%: number analyzed (Participants) | 72
  Weight - Decrease from baseline of >7% | 32

5. Secondary Outcome: Change in ALSFRS-R (ALS Functional Rating Scale With Respiratory Component) Total Score From Baseline to Week 12
Description: The ALSFRS-R (ALS functional rating scale with respiratory component) is a validated scale which measures 4 functional domains, comprising respiratory function, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48. Therefore, the score ranges from 0 to 48 with higher scores representing better function.
Time Frame: 12 weeks
Population: All subjects who received at least 1 dose of study treatment during the study and who at least one valid post-baseline measurement and a measurement at the timepoint being analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 69
units on a scale | -2.48 (3.424)

6. Secondary Outcome: Change in ALSFRS-R (ALS Functional Rating Scale With Respiratory Component) Total Score From Baseline to Week 24
Description: as for outcome 5
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 55
units on a scale | -4.29 (4.589)

7. Secondary Outcome: Change in ALSFRS-R (ALS Functional Rating Scale With Respiratory Component) Total Score From Baseline to Week 48
Description: as for outcome 5
Time Frame: 48 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 45
units on a scale | -7.49 (8.476)

8. Secondary Outcome: Change in Upright Vital Capacity From Baseline to Week 12
Description: Change in Percent Predicted Upright Vital Capacity from Baseline to Week 12. A negative change indicates clinical worsening.
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of predicted vital capacity
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 55
percentage of predicted vital capacity | -7.7 (14.03)

9. Secondary Outcome: Change in Upright Vital Capacity From Baseline to Week 24
Description: Change in Percent Predicted Upright Vital Capacity from Baseline to Week 24. A negative change indicates clinical worsening.
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of predicted vital capacity
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 48
percentage of predicted vital capacity | -12.5 (18.90)

10. Secondary Outcome: Change in Upright Vital Capacity From Baseline to Week 48
Description: Change in Percent Predicted Upright Vital Capacity from Baseline to Week 48. A negative change indicates clinical worsening.
Time Frame: 48 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of predicted vital capacity
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 35
percentage of predicted vital capacity | -15.8 (17.59)

11. Secondary Outcome: Change in McGill Single-Item Scale (SIS) From Baseline to Week 12
Description: The McGill SIS consists of a single question designed to assess the improvement of or the rate of deterioration of the subject's quality-of-life. Subjects rated their quality of life over the prior 2 days on a scale of 0 (very bad) to 10 (excellent). Decreases from Baseline indicate deterioration of a subject's quality of life.
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 69
units on a scale | -0.1 (1.48)

12. Secondary Outcome: Change in McGill Single-Item Scale (SIS) From Baseline to Week 24
Description: as for outcome 11
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 54
units on a scale | -0.5 (2.05)

13. Secondary Outcome: Change in McGill Single-Item Scale (SIS) From Baseline to Week 48
Description: as for outcome 11
Time Frame: 48 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 45
units on a scale | -0.8 (1.76)

14. Secondary Outcome: Number of Subjects With Feeding Tube Placed During the Study.
Description: Number of participants who had a feeding tube placed during the study.
Time Frame: 144 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical status evaluation. Subjects who had a feeding tube in place at the beginning of the study were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | KNS-760704 300 mg/Day
Number analyzed (Participants) | 70
participants | 24

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and reported from the first dose through 30 days following the last dose.
Arm/Group | 300 mg Per Day
All-Cause Mortality (participants affected / at risk) | 38/74
Serious Adverse Events (participants affected / at risk) | 48/74
Other Adverse Events (participants affected / at risk) | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg Per Day (N=74)
Neutropenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Oedema (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 5
Pyelonephritis acute (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Acinetobacter infection (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Face injury (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 25
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Wound drainage (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg Per Day (N=74)
Anaemia (Blood and lymphatic system disorders) | 5
Tachycardia (Cardiac disorders) | 6
Constipation (Gastrointestinal disorders) | 27
Salivary hypersecretion (Gastrointestinal disorders) | 17
Dysphagia (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 4
Ileus (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Oedema peripheral (General disorders) | 17
Fatigue (General disorders) | 11
Pyrexia (General disorders) | 13
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 7
Urinary tract infection (Infections and infestations) | 19
Bronchitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 10
Oral candidiasis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 6
Fall (Injury, poisoning and procedural complications) | 24
Contusion (Injury, poisoning and procedural complications) | 8
Procedural pain (Injury, poisoning and procedural complications) | 4
Weight decreased (Investigations) | 11
Blood triglycerides increased (Investigations) | 4
White blood cell count increased (Investigations) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Dysarthria (Nervous system disorders) | 13
Amyotrophic lateral sclerosis (Nervous system disorders) | 4
Headache (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 7
Urinary retention (Renal and urinary disorders) | 8
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes